CLINICAL TRIAL: NCT03554057
Title: Coronary Computed Tomographic Angiography to Optimize the Diagnostic Yield of Invasive Angiography in Lower Risk Patients
Brief Title: CCTA to Optimize the Diagnostic Yield of Invasive Angiography
Acronym: CarDIA
Status: Completed | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Hamilton Academic Health Sciences Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 4697
Record Dates: First submitted 2018-05-30; First posted 2018-06-12 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Coronary Artery Disease
Keywords: Angiogram, Coronary Computed Tomographic Angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group: All low-risk patients referred for invasive coronary angiography through the Hamilton General Hospital's Heart Investigation Unit Triage will be potentially eligible to receive the intervention over a 12-month period. The intervention will include risk stratification with CCTA at HHS and NHS as an alternative to upfront invasive angiography.
  Interventions: Diagnostic Test: Coronary Computed Tomographic Angiography
- Control Group: Intervention sites will act as their own controls: outcomes of all eligible patients in the 24-months prior to the implementation of the intervention will be assessed from a routinely collected health administrative database. Eligible patients not undergoing CCTA (patient or physician refusal, or CCTA not available) will be captured and included in the control group as part of a sensitivity analysis during the intervention period

INTERVENTIONS:
Diagnostic Test: Coronary Computed Tomographic Angiography — All low-risk patients referred for invasive coronary angiography will be potentially eligible to receive the intervention over a 12-month period. The intervention will include risk stratification using Coronary Computed Tomographic Angiography (CCTA) at HHS and NHS as an alternative to upfront invasive angiography. All CCTAs will be read by both a level 3-trained cardiologist and a radiologist. The results of the CCTA, coupled with evidence-based management recommendations will be sent to the referring physician and an invasive angiogram will be arranged only when indicated as per these management recommendations
  Groups: Intervention Group

SUMMARY:
This study aims to reduce patient risk and costs to the healthcare system by improving the diagnostic yield of invasive coronary angiography through existing triage processes to improve risk stratification using Coronary Computed Tomographic Angiography (CCTA) as a first step in low risk patients. All low-risk patients referred for invasive coronary angiography will be potentially eligible for CCTA instead of invasive angiography as a first-line diagnostic test. All CCTAs will be read by both a level 3-trained cardiologist and a radiologist. The results of the CCTA, coupled with evidence-based management recommendations will be sent to the referring physician and an invasive angiogram will be arranged by the HIU triage, only when clearly indicated

ELIGIBILITY:
Inclusion Criteria:

1. Non urgent outpatient referral
2. Canadian Cardiovascular Society class I or II
3. Indication for invasive angiogram includes: Rule out Coronary Artery Disease (CAD) and Cardiomyopathy

Exclusion Criteria:

1. Age <18 years old, Men >65 years old or women >75 years old
2. Patient refusal to provide verbal consent for CCTA at time of triage contact or unable to provide informed consent
3. Referring physician refusal for their eligible patients to be approached for the CarDIA study
4. Any prior CCTA
5. Atrial Fibrillation
6. Creatinine > 150 mmol/L
7. Diabetes mellitus
8. High risk Exercise Stress Test or Functional Imaging
9. Known severe valvular disease being considered for valve surgery
10. Any known CAD

    * Prior Acute Coronary Syndrome (ACS)
    * Prior Percutaneous Coronary Intervention (PCI) or Coronary Artery Bypass Graft (CABG)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible low-risk patients referred for invasive angiography will be recruited from the two interventional sites (approximately 240) via centralized triage process. Patients treated before the intervention implementation will be the control group (approximately 480).
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of invasive angiography | Three years
  Diagnostic yield is defined as the proportion of invasive angiograms that identify significant disease (≥70% stenosis) on a major coronary vessel (>2 mm) or > 50% stenosis in the left main)

SECONDARY OUTCOMES:
Quantitative assessment of angiograms avoided | Three years
  Number of angiograms avoided due to CCTA bookings
Deviation from management recommendations following CCTA | Three years
  Number of angiograms performed when not recommended
Protocol deviation as a surrogate for acceptability of the novel triage program | Three years
  Percentage of patients and physicians refusing to undergo CCTA as a first step
Costing of new strategy | Three years
  Cost of risk stratification of Coronary Artery Disease in low risk patients

CONTACTS AND LOCATIONS:
Overall Officials: Jon-David Schwalm, MD,FRCPC,Msc, Principal Investigator — Hamilton Health Sciences Corporation; Tej Sheth, Bsc,FRCPC,MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roth GA, Forouzanfar MH, Moran AE, Barber R, Nguyen G, Feigin VL, Naghavi M, Mensah GA, Murray CJ. Demographic and epidemiologic drivers of global cardiovascular mortality. N Engl J Med. 2015 Apr 2;372(14):1333-41. doi: 10.1056/NEJMoa1406656. PMID 25830423
- [Background] Sheth T, Amlani S, Ellins ML, Mehta S, Velianou J, Cappelli G, Yang S, Natarajan M. Computed tomographic coronary angiographic assessment of high-risk coronary anatomy in patients with suspected coronary artery disease and intermediate pretest probability. Am Heart J. 2008 May;155(5):918-23. doi: 10.1016/j.ahj.2007.11.035. Epub 2008 Feb 19. PMID 18440342
- [Background] Patel MR, Peterson ED, Dai D, Brennan JM, Redberg RF, Anderson HV, Brindis RG, Douglas PS. Low diagnostic yield of elective coronary angiography. N Engl J Med. 2010 Mar 11;362(10):886-95. doi: 10.1056/NEJMoa0907272. PMID 20220183
- [Background] Ouellette ML, Beller GA, Loffler AI, Workman VK, Bourque JM. Appropriate Referrals of Angiography Despite High Prevalence of Normal Coronary Arteries or Nonobstructive CAD. J Am Coll Cardiol. 2017 May 30;69(21):2673-2675. doi: 10.1016/j.jacc.2017.03.565. No abstract available. PMID 28545644
- [Background] Dewey M, Rief M, Martus P, Kendziora B, Feger S, Dreger H, Priem S, Knebel F, Bohm M, Schlattmann P, Hamm B, Schonenberger E, Laule M, Zimmermann E. Evaluation of computed tomography in patients with atypical angina or chest pain clinically referred for invasive coronary angiography: randomised controlled trial. BMJ. 2016 Oct 24;355:i5441. doi: 10.1136/bmj.i5441. PMID 27777234
- [Background] Zhang F, Wagner AK, Ross-Degnan D. Simulation-based power calculation for designing interrupted time series analyses of health policy interventions. J Clin Epidemiol. 2011 Nov;64(11):1252-61. doi: 10.1016/j.jclinepi.2011.02.007. PMID 21640554